CLINICAL TRIAL: NCT03849170
Title: Reducing Competitive Anxiety in Cheerleaders: A Psychological Approach
Brief Title: Reducing Competitive Anxiety Cheerleader Psychology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113455
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-01

CONDITIONS: Sports Injury; Stress Reaction; Performance Anxiety
Keywords: cheerleading; stress management; injury prevention; psychosocial factors; stress-injury; performance; coping skills; stress inoculation technique; competitive anxiety; psychological intervention
MeSH Terms: conditions — Athletic Injuries; Fractures, Stress | interventions — Play Therapy

STUDY DESIGN:
Intervention Model Description: Independent, randomized groups, longitudinal study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Intervention (Experimental): Six session intervention, each session 20-25 minutes in length. Stress inoculation technique-based intervention. Participants will be taught stress coping skills and relaxation skills such as self-efficacy statements, imagery, relaxation breathing, relaxation scripts, thought stoppage, cognitive reframing, positive self-talk, goal setting, event planning, and preparing for competition
  Interventions: Behavioral: Stress Inoculation Technique
- Health Intervention (Placebo Comparator): Six session intervention, each session 20-25 minutes in length. Participants will be taught relevant health and nutrition guidelines and practice using a food diary app (MyFitnessPal). Nutrition and health content will include such topics as reading Canadian food labels, vitamins and supplements, effects of alcohol on performance and recovery, vegetarian vs. omnivore diets, and hydration & performance.
  Interventions: Other: Health Intervention

INTERVENTIONS:
Behavioral: Stress Inoculation Technique — Teaches athletes to use cognitive-behavioral techniques to reduce their stress response during sporting events.
  Arms: Psychological Intervention
Other: Health Intervention — Will provide basic dietary and lifestyle guidelines that athletes should follow in their daily lives to maintain their health
  Arms: Health Intervention

SUMMARY:
Cheer leading is a rapidly growing international sport known for its acrobatic skills and dangerous stunts. The sport presents ample risk for physical trauma, and it is common for athletes to miss extensive time from cheer leading due to injury. The goal of this study is to the see whether the investigators can reduce injury risk among cheer leading athletes by teaching them stress-coping skills to help them relax and reduce their sport-related stress. There exists a link between high levels of stress and increased rates of injury among athletes. When individuals become stressed during athletic events such as competitions or strenuous training, symptoms including muscle tension and narrowed attention often accompany the stress response, increasing injury risk and reducing performance quality. In this study, half of Western University's coed cheer leading team will participate in a six-session stress management intervention to teach them relevant psychological stress-coping skills. Such skills include relaxation breathing techniques, visualization exercises, stoppage of negative thoughts, and development of self-efficacy statements. The other half of the team will receive a placebo "sport nutrition" program. The sessions of both the control program and the stress-management intervention will be administered over the most intensive period of the cheer leading season, from September to November of 2019. The investigators predict that the intervention group athletes will report less cheer leading time missed due to injury, report less sport-related stress, and make fewer errors at their cheer leading championship than their teammates in the placebo group. This is the first study to administer a psychological injury-prevention intervention to cheerleaders.

DETAILED DESCRIPTION:
Background Information: Cheer leading is a growing, highly competitive, and potentially stressful sport, with 3.5 million athletes practicing worldwide. The sport presents many risks, as it was responsible for more catastrophic injuries among female high school and college athletes than any other sport between 1982 and 2016 in the U.S. In Canada, there were 1496 cheer leading injuries requiring hospitalization from 1990 to 2010. According to the Williams and Andersen stress model, athletes with certain personality dispositions (e.g. high competitive anxiety), fewer coping resources (e.g. social support, stress management) and an extensive history of life stressors are prone to appraising athletic situations as being stressful, resulting in an exaggerated stress response. The stress response is particularly likely to manifest itself during instances in which an athlete perceives a high demand to succeed, but feels they possess inadequate resources to do so. These situations often lead to a variety of symptoms, including poorer performance quality, generalized muscle tension (physiological), and heightened distractibility (attentional), culminating in a greater likelihood of injury among athletes. Objectives: The goal of this study will be to administer a psychological-based intervention to improve the stress-coping skills of competitive cheerleaders, acting to minimize their competitive anxiety, maintain their performance quality, and reduce their risk of injury during the span of a season. Hypothesis: Cheerleaders who complete a psychological-based stress-coping intervention will report lower competitive anxiety, demonstrate superior performance, and report less time lost from cheer leading due to injury compared to a control group of teammates receiving a placebo program. Theoretical Approach: The psychological intervention will be based on the Stress Inoculation Technique (SIT), with the objective of restructuring athletes' coping skills in order to improve their management of stress (i.e. competitive anxiety). During the first phase of SIT, athletes will bring up narrative accounts of stressful athletic situations, identifying previously insufficient coping techniques as well as potential coping strengths. Self-monitoring strategies will be introduced to help athletes become more aware of the ways that they inadvertently build up stress reactions. During the second SIT phase, athletes will be taught coping skills such as muscle relaxation, use of self-efficacy (confidence) statements, cognitive re-framing of stressful situations, and emotion regulation techniques, which they will then apply to their personal cheer leading experiences. These skills will be further rehearsed through positive mental imagery and practice to ensure their effectiveness. In the final SIT stage, athletes will be encouraged to apply their new coping skills to incrementally more demanding cheer leading situations while utilizing stress management techniques. Athletes will be further reminded to take credit for their improvement, instilling a lasting sense of self-efficacy. The SIT intervention will teach athletes an array of anxiety management skills in order to help them develop effective stress-coping strategies during important cheer leading events. Participants will maintain an in-person correspondence with the researcher throughout to ensure a properly personalized and collaborative intervention experience. Methods: The intervention period will reach from September 2019 to December 2019, as this is the busiest and most competitive part of the cheer leading season. Half of Western University's 30-40 athlete co-ed cheer leading team will be randomized to complete a six session "sport nutrition" program as a control, while the other half will be randomized to complete a six session bi-weekly SIT program. Since the intervention and control groups will come from the same team, all participants will share identical practice and competition schedules, ensuring each group is exposed to the same athletic situations. As such, differences in group outcomes will most likely be due to the type of intervention they received. To measure performance quality, total scoring deductions caused by the athletes in each group during Western's two runs at the 2019 PCA college cheer leading championship will be compared. Fewer deductions indicate fewer errors (bobbles, drops, falls, etc.) and reflect superior performance. Impact: The current study will be the first to develop and implement a psychological-based intervention tailored to cheerleaders with the goal of improving these athletes' stress-coping abilities. If successful, this intervention is highly scalable and can be used by athletes where stress and injury are salient features of their sport, and where individual performance is highly scrutinized.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be active members of Western University's coed cheerleading team for the 2019 competitive season (August-November 2019)
* Participants must be on Western University's coed cheerleading team during the 2019 PCA College National Championships
* Participants must have no experience with psychological stress-management interventions aimed at reducing competitive sport anxiety, in particular, no previous experience with Stress Inoculation Technique therapy.

Exclusion Criteria:

* Not being an active member of Western University's coed cheerleading team for the beginning of the 2019 competitive season (September 2019), whether due to injury or absence from the team.
* Not being an active member of Western University's coed cheerleading team during the 2019 PCA College National Championships
* Previous experience with psychological stress-management interventions aimed at reducing competitive sport anxiety in a cheerleading context, in particular, previous experience with Stress Inoculation Technique therapy.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Injury Time | 14 weeks
  The amount of cheerleading time participants must modify or miss due to injuries suffered due to cheerleading. This outcome will be self-reported by each participant throughout the time frame using an injury data sheet provided to them by the investigators.
Incidences of Injury | 14 weeks
  The number of cheerleading injuries sustained by the participants during the study period. This outcome will be self-reported by each participant throughout the time frame using an injury data sheet provided to them by the investigators.

SECONDARY OUTCOMES:
Sport Anxiety | First at baseline, then again 14 weeks later.
  The amount of anxiety and stress participants report feeling as a result of the demands of training and competing for their cheerleading team. This outcome will be measured based on each participant's score on the Sport Anxiety Scale-2 (SAS-2). Each participant's post-test score on this measure will be compared to the participant's baseline score. There are fifteen questions, with five questions per subscale: somatic symptoms, concentration disruption, and worry. Each question asks participants how often they experience worry, concentration disruption, or somatic symptoms, with a low score of 1 indicating "not at all" and a high score of 4 indicating "very much". Total score on the questionnaire ranges from 15 to 60. A low total score indicates lower sports anxiety, and a higher scores indicates intense feelings of worry, disruption of concentration, and somatic symptoms.
Stress Coping Resources | First at baseline, then again 14 weeks later.
  The amount of stress coping techniques and skills participants employ in order to deal with their sport anxiety during important sporting events. This outcome will be measured based on each participant's score on the Athletic Coping Skills Inventory-28 (ACSI-28). Each participant's post-test score on this measure will be compared to the participant's baseline score. There are 28 questions, and seven subscales: coping with adversity, coachability, concentration, confidence and achievement motivation, goal-setting and mental preparation, peaking under pressure, and freedom from worry. Scores range from a low of 0 to a high of 12 on each subscale, with higher scores indicating greater strengths on that subscale. The score for the total scale ranges from a low of 0 to a high of 84, with higher scores signifying greater strength.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessis, Ph.D, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meichenbaum, D. H., & Deffenbacher, J. L. (1988). Stress Inoculation Training. The Counseling Psychologist, 16(1), 69-90.
- [Background] Williams, J. M., & Andersen, M. B. (1998). Psychosocial Antecedents of Sport Injury: Review and Critique of the Stress and Injury Model. Journal of Applied Sport Psychology, 10, 5-25.
- [Background] Smith, R. E., Schutz, R. W., Smoll, F. L., & Ptacek, J. T. (1995). Development and Validation of a Multidimensional Measure of Sport-Specific Psychological Skills: The Athletic Coping Skills Inventory-28. Journal of Sport and Exercise Psychology, 17, 379-398.
- [Background] Smith, R. E., Smoll, F. L., Cumming, S. P., & Grossbard, J. R. (2006). Measurement of Multidimensional Sport Performance Anxiety in Children and Adults: The Sport Anxiety Scale-2. Journal of Sport & Exercise Psychology, 28, 479-501.
- [Background] Hardy I, McFaull S, Saint-Vil D. Neck and spine injuries in Canadian cheerleaders: An increasing trend. J Pediatr Surg. 2015 May;50(5):790-2. doi: 10.1016/j.jpedsurg.2015.02.039. Epub 2015 Feb 19. PMID 25783366
- [Background] Kucera, K. L., Thomas, L. C., Cantu, R. C. (2017). Catastrophic Sports Injury Research, Thirty-Fourth Annual Report, Fall 1982 - Spring 2016. Chapel Hill, NC.
- [Result] Kolt GS, Hume PA, Smith P, Williams MM. Effects of a stress-management program on injury and stress of competitive gymnasts. Percept Mot Skills. 2004 Aug;99(1):195-207. doi: 10.2466/pms.99.1.195-207. PMID 15446646
- [Result] Maddison, R., & Prapavessis, H. (2005). A Psychological Approach to the Prediction and Prevention of Athletic Injury. Journal of Sport and Exercise Psychology, 27, 289- 310.